CLINICAL TRIAL: NCT03909633
Title: Effects of Intravenous Anesthesia on Postoperative Cognitive Function in Patients Accepted Painless Gastroenteroscopy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: IR2018001085
Record Dates: First submitted 2018-10-21; First posted 2019-04-10 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Postoperative Cognitive Function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A: anesthesia group: Patients accepting endoscopy check under anesthesia will be included in this group as group A,will doing a series of tests
  Interventions: Behavioral: a series of tests
- B:Non-anesthesia group: patients undergoing endoscopy check without anesthesia will be included in this group as controls voluntarily,namely group B,will doing a series of tests
  Interventions: Behavioral: a series of tests

INTERVENTIONS:
Behavioral: a series of tests — all patients in every group will do a series of tests,including DSST、DST、MoCA、WCST、HADS

SUMMARY:
The investigators want to study the effect of intravenous anesthesia on postoperative cognitive function in patients accepted gastroenteroscopy ,no additional medication or operation is involved

DETAILED DESCRIPTION:
The investigators want to study the effect of intravenous anesthesia on postoperative cognitive function in patients accepted gastroenteroscopy ,no additional medication or operation is involved.The investigators assess cognitive function through a series of tests for 4 times( within 3 days before the endoscopy ,2 hours after the endoscopy finished,1 week after the endoscopy,3 months after the endoscopy),including WCST、DSST、DST、HADS、MoCA,through self - contrast,the investigators will conclude whether intravenous anesthesia has bad impact on cognitive function or not .

ELIGIBILITY:
Inclusion Criteria:

* voluntary to participate in
* Vital signs are stable
* no drug or alcohol abuse
* no mental illness
* no severe central system diseases such as brain infarction
* between 18 and 80
* no liver or kidney dysfunction
* will perform endoscopy for various reasons

Exclusion Criteria:

* illiteracy
* color blindness
* can't write or refused to sign informed consent
* unable to follow up regularly or cooperate with the examination
* drug or alcohol abuse
* hearing or visual serious impairment
* has severe central nervous system diseases such as shoke ,neurosyphilis
* uncontrolled high blood pressure or hyperglycemia
* neurosyphilis
* history of craniotomy for various reasons
* liver and kidney dysfunction
* non-digestive tumors
* history of intravenous or general anesthesia for other causes in the last 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients will undergoing endoscopy check for all kinds of reasons
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in patient's cognitive dysfunction evaluated by WCST | 4 months
  The Wisconsin Card Sorting Test (WCST) is a neuropsychological test of "set-shifting",.A number of stimulus cards are presented to the participant. The participant is told to match the cards, but not how to match; however, he or she is told whether a particular match is right or wrong. The test takes approximately 12-20 minutes to carry out and generates a number of psychometric scores, including numbers, percentages, and percentiles of: categories achieved, trials, errors, and perseverative errors
Change in patient's cognitive dysfunction evaluated by DST | 4 months
  DST(Digit Span Test.),It is used to measure working memory's number storage capacity. Participants see or hear a sequence of numerical digits and are tasked to recall the sequence correctly, with increasingly longer sequences being tested in each trial. The participant's span is the longest number of sequential digits that can accurately be remembered. Digit-span tasks can be given forwards or backwards, meaning that once the sequence is presented, the participant is asked to either recall the sequence in normal or reverse order.Digit-span tasks are the most commonly used test for memory span, partially because performance on a digit-span task cannot be affected by factors such as semantics, frequency of appearance in daily life, complexity, etc.
Change in patient's cognitive dysfunction evaluated by DSST | 4 months
  DSST(Digit Symbol Test).,The participants need to write the number referred to each symbol in 90 seconds.Number of hits are registered. The test measures short-term memory, visualspatial skills and attention.
Change in patient's cognitive dysfunction evaluated by MoCA | 4 months
  MoCA （Montreal Cognitive Assessment）, The visual spatial executive ability, naming,memory, attention, language fluency, abstract,thinking, delayed memory and directional force are included in the test, a total of 30 points. The subjects whose have less than 12-year of education were added 1 point in the testing result, with correction of bias in the degree of culture. The patients whose get higher scores indicate that the cognitive function is better, 26 points as normal.

CONTACTS AND LOCATIONS:
Overall Officials: Cai J Ting, Study Chair — Second affiliated hospital of school of medicine, zhejiang university
Locations (1):
- Cai Jian Ting, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
to protect Patient privacy